CLINICAL TRIAL: NCT02012296
Title: A Phase I/II Trial of Enzalutamide Plus the Glucocorticoid Receptor Antagonist Mifepristone for Patients With Metastatic Castration Resistant Prostate Cancer (CRPC)
Brief Title: Enzalutamide and Mifepristone in Treating Patients With Metastatic Hormone Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-0979; NCI-2013-02151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDMRP-PC121149; IRB13-0979 (Other: University of Chicago); P30CA014599 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Results first posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Mifepristone

STUDY DESIGN:
Intervention Model Description: We report here the phase 2 results
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (enzalutamide) (Active Comparator): Patients receive enzalutamide PO per standard of care.
  Interventions: Drug: enzalutamide; Other: laboratory biomarker analysis; Other: pharmacological study
- Treatment (enzalutamide, mifepristone) (Experimental): Patients receive enzalutamide PO and mifepristone PO.
  Interventions: Drug: enzalutamide; Drug: mifepristone; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: enzalutamide — Given PO
  Other Names: MDV3100; selective androgen receptor modulator MDV3100; XTANDI
Drug: mifepristone — Given PO
  Other Names: Mifegyne; Mifeprex; RU-38486
  Arms: Treatment (enzalutamide, mifepristone)
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of enzalutamide and mifepristone when given together and to see how well they work in treating patients with metastatic hormone resistant prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as enzalutamide and mifepristone, may lessen the amount of androgens made by the body. It is not yet known whether enzalutamide is more effective with or without mifepristone in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safe and pharmacologically active doses of mifepristone and enzalutamide to use in combination. (Phase I) II. To determine if mifepristone in combination with enzalutamide prolongs time to prostate-specific antigen (PSA) progression compared to enzalutamide alone in patients with metastatic castration resistant prostate cancer. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the effect of mifepristone on endocrine biomarkers such as serum cortisol and thyrotropin.

II. To determine the effect of mifepristone on enzalutamide clearance and steady state enzalutamide exposure.

III. To determine if mifepristone affects PSA response rate when added to enzalutamide.

IV. To determine if mifepristone when added to mifepristone prolongs radiographic and clinical progression free survival according to standard working group criteria.

V. To explore the role of glucocorticoid receptor (GR) and androgen receptor (AR) protein expression within circulating tumor cells as a pharmacodynamic biomarker for mifepristone and enzalutamide in castration resistant prostate cancer (CRPC).

VI. To explore the expression of GR and down-stream AR/GR targets in metastatic tumor specimen prior to combination drug administration and at clinical progression.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

PHASE I: Patients receive enzalutamide orally (PO) on days 1-57 and mifepristone PO on days 29-57. Treatment continues in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive enzalutamide PO for 12 weeks per standard of care. Patients are then randomized to 1 of 2 treatment arms.

ARM I: Patients receive enzalutamide PO per standard of care.

ARM II: Patients receive enzalutamide PO and mifepristone PO.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer
* Evidence of castrate testosterone level < 50 ng/dL (or surgical castration)
* For Phase I portion of the study: evidence of disease progression:

  * 2 or more new lesions on bone scan or
  * Progressive disease on computed tomography (CT)/magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria or
  * Rising PSA: PSA evidence for progressive prostate cancer consists of a minimum PSA level of at least 2 ng/ml, which has subsequently risen on at least 2 successive occasions, at least 2 weeks apart
* For Phase II portion of the study:

  * Subjects must be on enzalutamide for metastatic CRPC and within the first 12 weeks of enzalutamide at 160mg/day
  * Record of subject's enzalutamide start date and baseline PSA (within 28 days of starting) before starting enzalutamide available
* Subjects must have documented clinically stable disease or better during the screening period of the study as defined by all of the following:

  * PSA =<1.25 times the PSA at start of enzalutamide
  * Lack of radiographic progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and Prostate Cancer Working Group Criteria
  * Clinically stable as confirmed by treating physician
* Any prior therapy for castrate disease is acceptable except prior specific cytochrome P450 family 17 (CYP17) antagonists (e.g. abiraterone acetate, orteronel) or prior second generation AR antagonists (e.g. enzalutamide or ARN509) which are excluded other than enzalutamide as specified for phase II portion; a minimum washout of 28 days for any other anticancer therapy prior to first dose of study drug is required (only applicable for phase I)
* Any other radiotherapy or radionuclide require 28-day washout prior to first dose of study drug
* Denosumab or zoledronic acid are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin =< 1.5 x the upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), finasteride (Proscar), dutasteride (Avodart), or any herbal product known to decrease PSA levels (e.g., saw palmetto and PC-SPES), or any systemic corticosteroid within 2 weeks prior to first dose of study drug
* Inability to swallow capsules or known gastrointestinal malabsorption
* History of other malignancies, with the exception of: adequately treated non-melanoma skin cancer, adequately treated superficial bladder cancer, stage 1 or 2 solid tumor malignancies who are without evidence of disease, or other solid tumors curatively treated with no evidence of disease for >= 5 years from enrollment
* Blood pressure that is not controlled despite > 2 oral agents (systolic blood pressure [SBP] > 160 and diastolic blood pressure [DBP] > 90 documented during the screening period with no subsequent blood pressure readings < 160/100)
* History of seizure disorder or active use of anticonvulsants
* Corrected QT interval (QTc) on electrocardiogram (EKG) > 450 msec
* Serious intercurrent infections or non-malignant medical illnesses that are uncontrolled
* Active psychiatric illness/social situations that would limit compliance with protocol requirements
* New York Heart Association (NYHA) class II, NYHA class III, or IV congestive heart failure (any symptomatic heart failure)
* Concurrent therapy with strong inhibitors or inducers of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) or cytochrome P450 family 2, subfamily C, polypeptide 8 (CYP2C8) due to concerning possible drug-drug interactions

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-12-13 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Szmulewitz, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois (Decatur) /Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Wayne State University Karmanos Cancer Institute, Detroit, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Enzalutamide): Patients receive enzalutamide 160 mg daily during a 12-week lead-in followed by enzalutamide 160 mg daily per standard of care.
  enzalutamide: Given PO
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Treatment (Enzalutamide, Mifepristone): Patients receive enzalutamide 160 mg daily during a 12-week lead-in followed by enzalutamide 120 mg daily plus mifepristone 300 mg daily.
  enzalutamide: Given PO
  mifepristone: Given PO
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Not Randomized: Patients received Enzalutamide 160 mg daily during a 12-week lead-in.
Period: Overall Study
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Started | 33 | 33 | 22
Completed | 33 | 32 | 0
Not Completed | 0 | 1 | 22
Not completed — Lack of Efficacy | 0 | 0 | 15
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Early study closure | 0 | 0 | 5
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Enzalutamide): Patients receive enzalutamide 160 mg daily during a 12-week lead-in followed by enzalutamide 160 mg daily per standard of care.
  enzalutamide: Given PO
- Treatment (Enzalutamide, Mifepristone): Patients receive enzalutamide 160 mg daily during a 12-week lead-in followed by enzalutamide 120 mg daily plus mifepristone 300 mg daily.
  enzalutamide: Given PO
  mifepristone: Given PO
- Total: Total of all reporting groups
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized | Total
Number analyzed (Participants) | 33 | 33 | 22 | 88
Age, Continuous [Median (Full Range); unit: years] | 71 [52 to 83] | 71 [57 to 85] | 68 [52 to 88] | 70 [52 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 33 | 33 | 22 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 3 | 19
  White | 20 | 26 | 16 | 62
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 22 | 66

OUTCOME MEASURES:

1. Primary Outcome: PSA Progression-free Survival
Description: PSA progression was defined as a PSA that is ≥1.25 times (25% increase) the PSA at randomization (week 12) and an absolute 5 ng/ml increase. PSA progression-free survival is PSA progression or death from any cause.
Time Frame: Up to 3 years, measured from randomization
Population: Patients not randomized were not evaluated for PSA progression-free survival.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Not Randomized: Received enzalutamide160 mg daily during a 12-week lead-in.
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 33 | 32 | 0
Months | 20.8 [8.3 to NA] — Upper confidence limit cannot be estimated due to insufficient number of participants with events. | 16.5 [8.4 to NA] — Upper confidence limit cannot be estimated due to insufficient number of participants with events. |
Statistical Analysis 1: Comparison: Treatment (Enzalutamide) vs Treatment (Enzalutamide, Mifepristone); Test type: Superiority; p = 0.83, Log Rank

2. Secondary Outcome: Radiographic PFS
Description: Radiographic progression or death from any cause.
Time Frame: Up to 3 years, measured from randomization
Population: Patients not randomized were not evaluated for radiographic progression-free survival.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Not Randomized: Received enzalutamide 160 mg daily during a 12-week lead-in.
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 33 | 32 | 0
Months | NA [8.4 to NA] — Median and upper confidence limit cannot be estimated due to insufficient number of participants with events | 16.5 [8.3 to NA] — Upper confidence limit cannot be estimated due to insufficient number of participants with events. |
Statistical Analysis 1: Comparison: Treatment (Enzalutamide) vs Treatment (Enzalutamide, Mifepristone); Test type: Superiority; p = 0.21, Log Rank

3. Secondary Outcome: Number of Participants With Positive AR Expression Within Circulating Tumor Cells (CTCs)
Description: Positive/negative classification with positive defined as a cytokeratin cell for whom there was an androgen receptor > 0
Time Frame: Week 12 (randomization)
Population: Number of patients with circulating tumor cells.
Measure: Count of Participants; unit: Participants
Groups:
- Not Randomized: Received enzalutamide 160 mg daily during 12-week lead-in.
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 23 | 13 | 6
Participants | 16 | 8 | 5

4. Secondary Outcome: Number of Participants With Positive GR Expression Within Circulating Tumor Cells (CTCs)
Description: Positive/negative classification with positive defined as a cytokeratin cell for whom there was an glucocorticoid receptor > 0
Time Frame: Week 12 (randomization)
Population: Patients with circulating tumor cells (CTCs).
Measure: Count of Participants; unit: Participants
Groups:
- Not Randomized: Patients received enzalutamide 160 mg daily during 12-week lead-in.
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 23 | 13 | 6
Participants | 17 | 8 | 5

5. Secondary Outcome: Testosterone
Description: Change from week 12 to week 16
Time Frame: 12 to 16 weeks
Population: 6 patients in the enzalutamide arm and 7 patients in the enzalutamide plus mifepristone arm had missing data. Patients not randomized were not evaluated for changes in testosterone.
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 27 | 25 | 0
ng/dL | 0.6 (1.2) | 21.0 (6.0) |
Statistical Analysis 1: Comparison: Treatment (Enzalutamide) vs Treatment (Enzalutamide, Mifepristone); Test type: Superiority; p = 0.0012, t-test, 2 sided

6. Secondary Outcome: Thyroid Stimulating Hormone
Description: Change in log(TSH) from week 12 to week 16
Time Frame: 12 to 16 weeks
Population: 13 patients in the enzalutamide arm and 2 patients in the enzalutamide plus mifepristone arm had missing data. Patients not randomized were not evaluated for changes in TSH.
Measure: Mean (Standard Error); unit: log(mcU/mL)
Groups:
- Not Randomized: Received enzalutamide 160 mg during 12-week lead-in.
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 20 | 30 | 0
log(mcU/mL) | -0.121 (0.037) | 0.306 (0.097) |
Statistical Analysis 1: Comparison: Treatment (Enzalutamide); Test type: Superiority; p < 0.0001, t-test, 2 sided

7. Secondary Outcome: Cortisol
Description: Change in log(Cortisol) from week 12 to week 16
Time Frame: 12 to 16 weeks
Population: 12 patients in the enzalutamide arm and 1 patient in the enzalutamide plus mifepristone arm had missing data. Patients not randomized were not evaluated for changes in cortisol.
Measure: Mean (Standard Error); unit: log(ug/dL)
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
Number analyzed (Participants) | 21 | 31 | 0
log(ug/dL) | 0.072 (0.126) | 0.733 (0.102) |
Statistical Analysis 1: Comparison: Treatment (Enzalutamide) vs Treatment (Enzalutamide, Mifepristone); Test type: Superiority; p = 0.0002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Treatment (Enzalutamide) | Treatment (Enzalutamide, Mifepristone) | Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/33 | 1/33 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/33 | 6/33 | 3/22
Other Adverse Events (participants affected / at risk) | 33/33 | 30/33 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzalutamide) (N=33) | Treatment (Enzalutamide, Mifepristone) (N=33) | Not Randomized (N=22)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
White blood cell decreased (Investigations) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzalutamide) (N=33) | Treatment (Enzalutamide, Mifepristone) (N=33) | Not Randomized (N=22)
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 2
Alkaline phosphatase increase (Investigations) | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 14 | 5
Anxiety (Psychiatric disorders) | 5 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 1
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blurred vision (Eye disorders) | 2 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Confusion (Psychiatric disorders) | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 13 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Depression (Psychiatric disorders) | 5 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 10 | 6 | 3
Dizziness (Nervous system disorders) | 6 | 6 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2
Edema limbs (General disorders) | 5 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 4 | 0
Fatigue (General disorders) | 25 | 27 | 14
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 9 | 1
Genital edema (Reproductive system and breast disorders) | 3 | 0 | 0
Headache (Nervous system disorders) | 5 | 6 | 2
Hematuria (Renal and urinary disorders) | 3 | 4 | 0
Hot flashes (Vascular disorders) | 19 | 15 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 3 | 1
Hypertension (Vascular disorders) | 5 | 6 | 2
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Memory impairment (Nervous system disorders) | 3 | 4 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Nausea (General disorders) | 6 | 6 | 3
Pain (General disorders) | 10 | 9 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4 | 4
Platelet count decreased (Investigations) | 3 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 2 | 1
Renal calculi (Renal and urinary disorders) | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 4 | 4 | 0
Urinary incontinence (Renal and urinary disorders) | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 2 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Flu like symptoms (General disorders) | 0 | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
General disorders and administration site conditions - Other (General disorders) | 1 | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Investigations - Other (Investigations) | 0 | 2 | 0
Paresthesia (Nervous system disorders) | 0 | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 3 | 2
Upper respiratory infection (Infections and infestations) | 1 | 5 | 4
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0
Watering eyes (Eye disorders) | 0 | 2 | 0
Weight gain (Investigations) | 1 | 2 | 0
Weight loss (Investigations) | 0 | 5 | 2
White blood cell decreased (Investigations) | 0 | 2 | 0
Skin infection (Infections and infestations) | 1 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT02012296/Prot_SAP_000.pdf